CLINICAL TRIAL: NCT05790603
Title: Effect of Patent Hemostatic Device (PHD) With Quantitative Pressure on Radial Artery Hemostasis After CAG/PCI：a Randomized Controlled Trial
Brief Title: Effect of Patent Hemostatic Device (PHD) With Quantitative Pressure on Radial Artery Hemostasis After CAG/PCI
Acronym: PCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023SF05
Record Dates: First submitted 2023-02-22; First posted 2023-03-30 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Coronary Intervention; Hemostasis
Keywords: Percutaneous coronary intervention; Radial artery hemostasis; Quantitative pressure; Randomized controlled trial
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: One of the primary outcome of radial artery occlusion will be assessed by masking the assessor. The data analyzers will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): PHD-band Group
  Interventions: Device: Intervention group with PHD-Band
- Control group (Active Comparator): TR-band Group
  Interventions: Device: Control group with TR-Band

INTERVENTIONS:
Device: Intervention group with PHD-Band — The initial compression pressure was systolic blood pressure plus 10mmHg. Pressure will be released by 20mmHg and 40mmHg 1 hour and 2 hours respectively after the surgery and then the band will be removed after 3 hours if no bleeding occurs. The compression will continue if bleeding occurs.
  Other Names: Brand name: WEGO Medical Products Group CO. LTD, China
  Arms: Intervention group
Device: Control group with TR-Band — TR-Band will be inflated with 15 mL of air The band will be deflated with 1 mL of air hourly for the following 2 hours after the procedure. After 3 hours, the band will be removed if no bleeding occurs. If rebleeding occurs, the band will be inflated with appropriate volume of air until bleeding stops .
  Other Names: Brand name: Terumo Medical Corporation, Japan
  Arms: Control group

SUMMARY:
The objective of this clinical trial is to compare the hemostatic effect of 2 hemostatic devices with or without quantitative pressure on radial arteries after coronary angiography (CAG) or percutaneous coronary intervention (PCI). The main questions aims to answer:

* What is the hemostatic effect of the patent hemostatic device with quantitative pressure after percutaneous coronary intervention?
* What are the precise hemostatic pressure and hemostatic time of the radial artery after CAG/PCI? Participants will be randomly assigned to the intervention group (IG) and control group (CG). The IG will use patent hemostatic device with quantitative pressure (PHDQP-Band, China) while the CG will use the conventional radial artery hemostatic device (TR-Band, Japan) without pressure monitoring.

The primary outcomes is incidence of 24h radial artery occlusion (24h RAO). Secondary outcomes include time to hemostasis, bleeding, hematoma, 30d radial artery occlusion (30d RAO), pain, hand swelling, numberness, pseudoaneurysm, and radial artery stenosis.

DETAILED DESCRIPTION:
The objective of this clinical trial is to compare the hemostatic effect of 2 hemostatic devices with or without quantitative pressure on radial arteries after percutaneous coronary intervention. The main questions aims to answer:

* What is the hemostatic effect of the patent hemostatic device after percutaneous coronary intervention?
* What are the precise hemostasis pressure and hemostasis time of the radial artery after percutaneous coronary intervention?

Participants will be randomly assigned to the intervention group (IG) and control group (CG).

For the participants assigned to the IG, the radial systolic pressure will be measured after TRA procedure. The PHD-Band with quantitative pressure ( WEGO Medical Products Group CO. LTD, China) will be placed at the entry site of the sheath. Connecting the hemostatic devices to the electric pneumatic machine with a connecting cable. After removing the radial sheath, the puncture site will be compressed by operator's hand. The PHD-Band with quantitative pressure will be inflated with specific pressure radial systolic pressure plus 10mmHg) and the hand will slowly release the pressure. If bleeding occurs, the PHD-Band will be deflated with 5-10mmHg automatically by parameter setting with the electric pneumatic machine until the bleeding stops. The PHD-Band will be deflated with20 mmHg, 40 mmHg of decreased pressure following 1h and 2h after the procedure. After 3 hours, the hemostatic pressure will be released to 45mmHg and the PHD-Band will be removed if no bleeding occurs. If rebleeding occurs, the band will be inflated according to the previous pressure for another an hour until bleeding stops.

For the participants assigned to the CG, the TR-Band (Terumo Medical Corporation, Japan) will be placed at the entry site of the sheath after TRA procedure and inflated with 10 mL of air and the radial sheath will be removed with hand compression. Another 5 mL of air will be inflated and the operator's hand will slowly release the pressure. The TR band will be inflated until bleeding stopped with the maximum air volume no more than 18ml. The band will be deflated with 1 mL of air hourly for the following 2 hours after the procedure. After 3 hours, the band will be deflated with 4 mL of air first and then all volume of the rest air if no bleeding occurs and then the band will be removed if no bleeding occurs. If rebleeding occurs, the band will be inflated with 1 mL of air until bleeding stops .

For all enrolled participants, the investigators will record the complications such as bleeding, subcutaneous hematoma, pain, hand swelling, numbness, pseudoaneurysm after the operation. Radial artery occlusion, subcutaneous hematoma, pseudoaneurysm, and radial artery stenosis were confirmed by arterial ultrasound within 24 hours and 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing coronary angiography or percutaneous coronary intervention via the radial artery; Positive Allen's test result; Willing to sign informed consent.

Exclusion Criteria:

Radial artery malformation； Chronic kidney disease with eGFR<30ml/min.1.73m2; Cirrhosis of the liver; Coagulation disfunction; Patients treated with IIb / IIIa receptor antagonist.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence early radial artery occlusion | Within 24 hours after CAG/PCI
  RAO occurs within 24 hours after CAG/PCI

SECONDARY OUTCOMES:
Compression time | through hemostasis completion，estimated to be an average of 3~6hours
  The interval from the time of sheath removal to the time of hemostasis removal
Incidence of access site bleeding | Within 24 hours after CAG/PCI
  Access site bleeding within 24 hours after CAG/PCI
Incidence of hematoma | through hemostasis completion，estimated to be an average of 4~6hours
  The incidence of subcutaneous hematoma in the distal skin of the compression site 24 h after the removal of the compression device
Incidence of 30d radial artery occlusion | Within 30 days after CAG/PCI
  RAO occurs within 30 days after CAG/PCI
The degree of pain | baseline; 24 hours after PCI
  Pain level is classified as painless: 0; mild pain: 1~3; moderate pain: 4~6; severe pain: 7~10.
numbness | baseline; 24 hours after PCI
  Numbness level is classified as no numbness with 0, mild numbness: 1~2; moderate numbness: 3; severe numbness:4~5
Hand swelling | baseline; 24 hours after PCI
  The circumference diameter of both hands was measured using a tape gauge contrast.
pseudoaneurysm | Within 24 hours after PCI
  It refers to the lumen of the same as the artery formed by the blood through the perivascular tissue after arterial puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhui Tao, Study Chair — Peking University First Hospital
Locations (2):
- China (2):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petroglou D, Didagelos M, Chalikias G, Tziakas D, Tsigkas G, Hahalis G, Koutouzis M, Ntatsios A, Tsiafoutis I, Hamilos M, Kouparanis A, Konstantinidis N, Sofidis G, Pancholy SB, Karvounis H, Bertrand OF, Ziakas A. Manual Versus Mechanical Compression of the Radial Artery After Transradial Coronary Angiography: The MEMORY Multicenter Randomized Trial. JACC Cardiovasc Interv. 2018 Jun 11;11(11):1050-1058. doi: 10.1016/j.jcin.2018.03.042. PMID 29880098
- [Background] Deitrich-MacLean G, Walden T. Distinguishing teaching interactions of physically abusive from nonabusive parent-child dyads. Child Abuse Negl. 1988;12(4):469-79. doi: 10.1016/0145-2134(88)90064-6. PMID 3233513
- [Background] Kulyassa P, Nemeth BT, Ehrenberger R, Ruzsa Z, Szuk T, Fehervari P, Engh MA, Becker D, Merkely B, Edes IF. The Design and Feasibility of the: Radial Artery Puncture Hemostasis Evaluation - RAPHE Study, a Prospective, Randomized, Multicenter Clinical Trial. Front Cardiovasc Med. 2022 May 27;9:881266. doi: 10.3389/fcvm.2022.881266. eCollection 2022. PMID 35694680
- [Result] Eid-Lidt G, Reyes-Carrera J, Farjat-Pasos JI, Saenz AL, Bravo CA, Rangel SN, Salido DZ, Vega Servin NS, Soto-Lopez ME, Gaspar J. Prevention of Radial Artery Occlusion of 3 Hemostatic Methods in Transradial Intervention for Coronary Angiography. JACC Cardiovasc Interv. 2022 May 23;15(10):1022-1029. doi: 10.1016/j.jcin.2022.03.011. PMID 35589232